CLINICAL TRIAL: NCT03091621
Title: Japanese Registry of Rivaroxaban Effectiveness & Safety for the Prevention of Recurrence in Patients With Deep Vein Thrombosis and Pulmonary Embolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nihon University (Other)
Collaborators: Mebix Inc (Industry)
Responsible Party: Principal Investigator, Atsushi Hirayama, Principal Investigator, Nihon University School of Medicine Division of Cardiology, Department of Internal Medicine, Nihon University
Other Study IDs: J'xactly
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Deep Vein Thrombosis; pulmonary embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To clarify the effectiveness and safety of the direct factor Xa inhibitor rivaroxaban in domestic clinical use for patients with deep vein thrombosis and pulmonary embolism

DETAILED DESCRIPTION:
Research design: multicenter collaboration, prospective, non-interventional, observational research

Research outline:

Registration period: Dec 2016 (after ethics committee approval) to May 2018 (1 year and 6 months) Investigation period: Dec 2016 (after ethics committee approval) to Nov 2019 (At least 1 year and 6 months) Target number of participants: 1,000 participants Estimated number of participating institutions: 150 medical institutions Research secretariat: Mebix, Inc.

Research procedure:

* Perform patient registration within 3 weeks of first prescription
* Also record when the drug was discontinued for any reason, such as an event or bleeding etc, between the time of first prescription and registration
* Track progress as much as possible until the end of the study period, regardless of continuation or discontinuation of study drug administration, and also in cases where there is manifestation of efficacy or safety events
* Track progress of all cases as much as possible until the end of the study period, regardless of continuation, discontinuation or termination of study drug administration. Patients transferred to the hospital are managed in the same way.

Registration method:

Register case information in the WEB registration system (EDC) after obtaining written consent from the research participant him/herself or the legal guardian for all cases compliant with the registration criteria and not in conflict with the exclusion criteria. Administer rivaroxaban in compliance with the approved dosage in the separate attached document. Furthermore, when the usage or dose are adjusted at the discretion of the research doctor, record the dose adjustment and reason. EDC will be used for case data entry.

[EDC; Items to be entered into the case registration screen]

1. Registration date
2. Facility name
3. Case registration number
4. Patient identification code (appropriate number within the facility)
5. Gender
6. Birthdate
7. Rivaroxaban commencement date
8. Age at first prescription (automatic calculation display)
9. Date of obtaining written consent
10. Other

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic or asymptomatic venous thromboembolism prescribed rivaroxaban

Exclusion Criteria:

1. Contraindication to rivaroxaban
2. Chronic thromboembolic pulmonary hypertension (however, it is possible to register if there is coexisting acute pulmonary embolism or deep vein thrombosis)
3. Active bleeding
4. Patients determined to be inappropriate for the study by the attending doctor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic or asymptomatic venous thromboembolism prescribed rivaroxaban for the purpose of treatment and prevention of recurrence of acute deep vein thrombosis and pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence/exacerbation of symptomatic venous thromboembolism (VTE) | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)

SECONDARY OUTCOMES:
Onset/exacerbation of symptomatic pulmonary embolism (PE) | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Onset/exacerbation of symptomatic deep vein thrombosis (DVT) | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Major bleeding event (ISTH bleeding criteria) | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Non-major bleeding event (bleeding events that do not correspond to major bleeding) | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Recurrence/exacerbation of symptomatic venous thromboembolism during the initial strengthening treatment period | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Bleeding event during the initial strengthening treatment period | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Acute coronary syndrome | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Cerebral infarction | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
VTE related death | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Cardiovascular death | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
All deaths | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Relationship between change in D-dimer and recurrence | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Comparison of examples of treatment continuation/discontinuation events | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)
Serious adverse events | From the time of research participation to 30th November 2019 (At least 1 year and 6 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Nihon University School of Medicine, Tokyo, Itabashi-ku, Japan

REFERENCES:
- [Derived] Okumura Y, Fukuda I, Nakamura M, Yamada N, Takayama M, Maeda H, Yamashita T, Ikeda T, Mo M, Yamazaki T, Hirayama A; J'xactly Investigators. Design and rationale for the Japanese Registry of Rivaroxaban Effectiveness & Safety for the Prevention of Recurrence in Patients with Deep Vein Thrombosis and Pulmonary Embolism (J'xactly) study. BMJ Open. 2018 Jun 22;8(6):e020286. doi: 10.1136/bmjopen-2017-020286. PMID 29934383